CLINICAL TRIAL: NCT02056548
Title: Comparison of the Occurrence of HBV Reactivation According to the Duration of Preemptive Antiviral Therapy in Chronic Hepatitis B Virus Carriers Receiving Cancer Chemotherapy for Hematologic Diseases
Brief Title: Hepatitis B Virus Reactivation After Withdrawal of Preemptive Antiviral Therapy in Hematologic Malignancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Jae-Ho, Yoon, Clinical fellowship in Catholic BMT Center, Seoul St. Mary's Hospital
Other Study IDs: CHSCTC-R01-HEPATO
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma; Chronic Hepatitis B
Keywords: preemptive antiviral treatment; lymphoma; chronic hepatitis B
MeSH Terms: conditions — Lymphoma; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Previous studies dealt with patients who maintained antiviral drugs for 2 ~ 6 months after final chemotherapy and they revealed that many of the patients who stopped preemptive antiviral drug within 6 months experienced viral reactivation. Based on the study results, guidelines recommend that preemptive antiviral therapy should be maintained for at least 6 months. Nevertheless, many clinicians apply the preemptive antiviral drugs for 1~2 years or longer after final chemotherapy without definite evidences, and this practice increases the medical expenditure a lot. Therefore, the investigators are going to find out the proper and safe duration of preemptive antiviral therapy which can be a good reference in the future practice.

DETAILED DESCRIPTION:
HBV reactivation in cancer patients is important not only for directly affecting severe hepatic failure but also for delaying of the further cancer treatments which may cause reduction of overall survival. Thus the guidelines according to the previous studies and other follow-up of randomized studies revealed that patients with positive HbsAg should be administered with preemptive antiviral therapy at least 6 month or more.

However, ideal duration for preemptive antiviral therapy to suppress viral reactivation and withdrawal hepatitis is not clearly identified at present time. It is because previous data just dealt with the efficiency of preemptive antiviral therapy, but most of them did not analyze the outcomes after withdrawal of antiviral therapy. Frequent late-onset reactivation hepatitis in association with preemptive antiviral therapy is mainly due to drug-resistance or post-withdrawal manifestation. Drug-resistance was mainly associated with lamivudine which is now substituted by entecavir or tenofovir which produce lower incidence of resistance (< 1.2% at 6 years). Therefore, the only issue at present is withdrawal hepatitis which may be due to early cessation of the antiviral drug.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* ECOG performance status 0, 1, 2
* Hodgkin's or Non-Hodgkins lymphomas according to the WHO 2008 classification
* Patients who received standard cytotoxic chemotherapies
* Patients who finished chemotherapy (duration not exceeded 6 months) or who will finish the planned chemotherapy
* Patients who achieved at least partial response and do not need further chemotherapy
* HBsAg (+) patients who received preemptive antiviral therapies

Exclusion Criteria:

* Anti-HCV Ab(+), HIV(+), or autoimmune hepatitis
* Complications due to uncompensated liver cirrhosis
* Child pugh score : 10 points or more
* Hepatocellular carcinoma
* Patients who finish the lymphoma treatments with only radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients who will be newly diagnosed as malignant lymphomas and receive standard chemotherapies at Seoul St. Mary's Hospital in Korea.
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of hepatitis B viral reactivation | within one year after cessation of the antiviral drug

SECONDARY OUTCOMES:
Severity of reactivation of hepatitis B | within one year after cessation of anviral drugs
  Severity according to ALT (IU/L) level Mild : up to 5 times from upper normal limit Moderate : 5- 10 times from upper normal limit Severe : ALT > 300 IU/L or ≥ 10 times